CLINICAL TRIAL: NCT00176098
Title: Correlation of Stress, Patient Comfort and Safety to Bispectral Index in Patients Under Hypnosis for Cataract Surgery
Brief Title: Hypnosis for Eye Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TF-KliMa-2005-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-02-07 (Estimated); Status verified 2005-09

CONDITIONS: Cataract
Keywords: Cataract surgery; Hypnosis; C11.510.245; F04.754.424.771; Suggestion
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Procedure: Hypnoanalgesia; Hypnotic shielding

SUMMARY:
Perioperative stress for cataract surgery in the elderly is considerable even in the absence of pain. For these patients with a high comorbidity level, the perioperative situation comprising factors such as uncomfortable positioning, dull ambience, face cover, poor sedation, and anxiety might not only reduce intraoperative compliance but induce cardiac ischemia and hypertensive crises. Hypnosis is supposed to increase patient comfort, to shield the patient from organic stress and to improve intraoperative compliance without side effects even in old and very ill patients. In a controlled study, we, the investigators at the University of Heidelberg, compared phakoemulsification under topical anesthesia as usual (and placebo hypnosis) with either additional hypnosis or hypnoanalgesia without topical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Cataract

Exclusion Criteria:

* Uncorrected hearing disability
* Pharmacological beta-blockade

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2005-09

PRIMARY OUTCOMES:
Reduction of perioperative stress
Improvement of patient comfort and safety

SECONDARY OUTCOMES:
Correlation of hypnotic depth with bispectral index (BIS)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, MD, PhD, Study Chair — Dept. of Anesthesiology and Critical Care Medicine, Faculty of Clinical Medicine Mannheim, University of Heidelberg
Locations (1):
- Dept. of Anesthesiology and Critical Care Medicine, Faculty of Clinical Medicine Mannheim, University of Heidelberg, Mannheim, Germany